CLINICAL TRIAL: NCT04073693
Title: Characterization of the Nutritional Status in the Patient With Liver Cirrhosis and Impact of a Nutritional Intervention With Nutritional Supplements With BRCA vs. Standard Treatment in the Subgroup of Patients With Sarcopenia
Brief Title: Characterization of the Nutritional Status in the Patient With Liver Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Jose Luis Calleja, Director. Clinical Research, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11.17
Record Dates: First submitted 2019-08-09; First posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Amino Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BRCA (Active Comparator): They were in treatment with BRCA and standard treatment based on nutritional intervention and physical exercise.
  Interventions: Dietary Supplement: Branched chain amino acids (BRCA)
- Placebo (Placebo Comparator): They only were on standard treatment based on nutritional intervention and physical exercise.
  Interventions: Dietary Supplement: Branched chain amino acids (BRCA)

INTERVENTIONS:
Dietary Supplement: Branched chain amino acids (BRCA) — They were with BRCA during the day apart of following the standard recommendations

SUMMARY:
In the subgroup of patients with sarcopenia, regardless of their body mass index, we want to verify the real impact of nutritional supplements with branched chain amino acids on the standard treatment based on nutritional intervention and physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients with sarcopenia in abdominal CT.

Exclusion Criteria:

* chronic renal failure or being on hemodialysis
* active hepatitis B or C virus infection
* active alcohol abuse
* coinfection with human immunodeficiency virus
* renal or previous liver transplantation
* history of neoplasia requiring chemotherapy or radiotherapy
* hepatocellular carcinoma outside of Milan criteria
* TIPs
* unwillingness to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Change of muscle mass in patients with sarcopenia | 12 weeks
  To assess whether to add to dietary and physical activity recommendations, nutritional supplements with BRCA under usual clinical conditions can lead to a greater change of muscle mass in patients with sarcopenia

CONTACTS AND LOCATIONS:
Locations (1):
- Jose Luis Calleja, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hernandez-Conde M, Llop E, Gomez-Pimpollo L, Fernandez Carrillo C, Rodriguez L, Van Den Brule E, Perello C, Lopez-Gomez M, Abad J, Martinez-Porras JL, Fernandez-Puga N, Ferre C, Trapero M, Fraga E, Calleja JL. Adding Branched-Chain Amino Acids to an Enhanced Standard-of-Care Treatment Improves Muscle Mass of Cirrhotic Patients With Sarcopenia: A Placebo-Controlled Trial. Am J Gastroenterol. 2021 Nov 1;116(11):2241-2249. doi: 10.14309/ajg.0000000000001301. PMID 34074812